CLINICAL TRIAL: NCT01995734
Title: An ACromegaly, Open-label, Multi-CEnter, Safety Monitoring Program for Treating Patients With SOM230 (Pasireotide) LAR Who Have Need to Receive Medical Therapy (ACCESS)
Brief Title: An Open-label, Multi-center, Expanded Treatment Protocol of Pasireotide LAR in Patients With Acromegaly
Acronym: ACCESS
Status: Approved for marketing | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CSOM230CUS33
Record Dates: First submitted 2013-11-20; First posted 2013-11-27 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Acromegaly
Keywords: Acromegaly, Pituitary diseases
MeSH Terms: conditions — Acromegaly; Pituitary Diseases

INTERVENTIONS:
Drug: Pasireotide long acting release formulation — Pasireotide LAR will be administered intramuscularly (i.m.) every 28 days until pasireotide becomes commercially available and reimbursed or until 31 December 2015, whichever occurs first.
  Other Names: SOM230 LAR

SUMMARY:
The present study is planned as an expanded treatment protocol to provide acromegalic patients for whom medical therapy is appropriate access to pasireotide LAR while regulatory approval for pasireotide is sought.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of active acromegaly with elevated IGF-1 (>ULN) and random GH (>1 μg/L) within 30 days of screening.
* Patients who are not controlled by pituitary surgery or who are not eligible for or refuse surgery.
* For patients on medical treatment for acromegaly the following washout periods must be completed before screening assessments are performed:

  * Dopamine agonists (bromocriptine, cabergoline): 4 weeks
  * GH-receptor antagonists (pegvisomant): 8 weeks
  * Somatostatin analogues: no washout period required
* Karnofsky performance status ≥ 60.

Exclusion Criteria:

* Concomitant treatment with somatostatin analogues unless concomitant treatment was discontinued 28 days before first pasireotide LAR injection is administrated.
* Concomitant treatment with growth hormone receptor (GHR)-antagonists or dopamine agonists unless concomitant treatment was discontinued and the washout period was completed before the screening assessments are performed.
* Patients with compression of the optic chiasm causing any visual field defect for whom surgical intervention is indicated.
* Patients who require a surgical intervention for relief of any sign or symptom associated with tumor compression.
* Patients who have undergone major surgery/surgical therapy for any cause within 4 weeks of screening.
* Patients who have received radiotherapy of the pituitary within 4 weeks prior to screening or have not recovered from side effects of radiotherapy.
* Patients who have a history of hypothyroidism and who are not adequately treated with stable doses of thyroid hormone replacement therapy.
* Patients with active malignant disease within the last five years (with the exception of basal cell carcinoma or carcinoma in situ of the cervix).
* Diabetic patients whose blood glucose is poorly controlled.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- United States (37):
  - University of Alabama at Birmingham Univ. of Alabama Birmingham, Birmingham, Alabama
  - Advanced Research, LLC Advanced Reserch (4), Peoria, Arizona
  - St. Joseph's Hospital Medical Center St. Joseph's Hosp Med Ctr (2), Phoenix, Arizona
  - San Diego Coastal Endocrinology Group, Chula Vista, California
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - University of California at Los Angeles UCLA - Los Angeles, Los Angeles, California
  - John Wayne Cancer Institute Saint John's Health Center, Santa Monica, California
  - Harbor-UCLA Medical Center Center for Men's Health, Torrance, California
  - George Washington University Medical Center Medical Faculty Associates Inc, Washington D.C., District of Columbia
  - Center for Diabetes & Endocrine Care Dept.of Ctr for Diab&Endoc - 2, Hollywood, Florida
  - Central Florida Endocrine & Diabetes Consultants, Maitland, Florida
  - Endocrine Assoc of FL, Ocoee, Florida
  - Emory University School of Medicine/Winship Cancer Institute Emory University (5), Atlanta, Georgia
  - Dr. Steven Leichter, Endocrine Consultant, Columbus, Georgia
  - Northwestern University Endo, Metabolism and Molecular, Chicago, Illinois
  - The Johns Hopkins University School of Medicine Johns Hopkins University, Baltimore, Maryland
  - Sinai Hospital of Baltimore Sinai Hospital, Baltimore, Baltimore, Maryland
  - Tufts Medical Center Tufts Medical Ctr, Boston, Massachusetts
  - Mayo Clinic - Rochester Mayo Clinic (2), Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - PALM MEDICAL RESEARCH CENTER Palm Research Center, Inc, Las Vegas, Nevada
  - Robert Wood Johnson Medical School Div. Endo, Meta & Nutrition, New Brunswick, New Jersey
  - University of New Mexico School of Medicine Univ of NM, Albuquerque, New Mexico
  - Stony Brook Internists PC, East Setauket, New York
  - Mount Sinai School of Medicine Mt. Sinai Schoof of Med., New York, New York
  - Columbia University Medical Center- New York Presbyterian Neuroendocrine Unit, New York, New York
  - Endocrine Associates of Long Island, P.C., Smithtown, New York
  - Endocrinology Associates Inc, Columbus, Ohio
  - Toledo Clinic Toledo Clinic, Inc., Toledo, Ohio
  - Oregon Health & Sciences University Oregon Health & Sciences, Portland, Oregon
  - Thomas Jefferson University Jefferson University Physician, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates Allegheny Endo Associates, Pittsburgh, Pennsylvania
  - MidState Endocrine Associates, Nashville, Tennessee
  - Vanderbilt University Medical Center Clinical Trials Center, Nashville, Tennessee
  - Baylor College of Medicine Division of Endocrinology, Houston, Texas
  - Virginia Endocrinology Research, Chesapeake, Virginia
  - Swedish Cancer Institute Swedish Neuroscience Institute, Seattle, Washington

REFERENCES:
- [Derived] Jerkins TW, Jerkins RK, Franklin R. Successful debulking of plurihormonal pituitary macroadenoma with long-acting pasireotide and dopamine agonist combination therapy. Clin Case Rep. 2019 Jan 28;7(3):445-451. doi: 10.1002/ccr3.1961. eCollection 2019 Mar. PMID 30899469
- [Derived] Lovato CM, Kapsner PL. Analgesic effect of long-acting somatostatin receptor agonist pasireotide in a patient with acromegaly and intractable headaches. BMJ Case Rep. 2018 Jun 19;2018:bcr2017219686. doi: 10.1136/bcr-2017-219686. PMID 29925553
- [Derived] Gordon MB, Nakhle S, Ludlam WH. Patients with Acromegaly Presenting with Colon Cancer: A Case Series. Case Rep Endocrinol. 2016;2016:5156295. doi: 10.1155/2016/5156295. Epub 2016 Nov 29. PMID 28025627
- [Derived] Fleseriu M, Rusch E, Geer EB; ACCESS Study Investigators. Safety and tolerability of pasireotide long-acting release in acromegaly-results from the acromegaly, open-label, multicenter, safety monitoring program for treating patients who have a need to receive medical therapy (ACCESS) study. Endocrine. 2017 Jan;55(1):247-255. doi: 10.1007/s12020-016-1182-4. Epub 2016 Nov 28. PMID 27896545